CLINICAL TRIAL: NCT02799888
Title: Safety and Efficacy of Maraviroc-Based Graft-Versus-Host-Disease Prophylaxis in HLA-Unrelated and HLA-Mismatched Related Donor Transplantation
Brief Title: Maraviroc-Based GVHD Prophylaxis in HLA-Unrelated and HLA-Mismatched Related Transplantation
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Affiliated Hospital to Academy of Military Medical Sciences (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 307-maraviroc-001
Record Dates: First submitted 2016-06-03; First posted 2016-06-15 (Estimated); Last update posted 2016-06-15 (Estimated); Status verified 2016-06

CONDITIONS: Graft-versus-host Disease; Hematopoietic Stem Cell Transplantation
Keywords: Graft-versus-host Disease; Hematopoietic Stem Cell Transplantation; Acute Leukemia; Myelodysplastic syndrome; Lymphoma
MeSH Terms: conditions — Graft vs Host Disease; Myelodysplastic Syndromes; Lymphoma | interventions — Maraviroc; Cyclosporine; Cyclosporins; Tacrolimus; Methotrexate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Maraviroc + standard GVHD prophylaxis (Experimental): Maraviroc administration (in addition to the standard prophylaxis therapy of cyclosporine/tacrolimus and methotrexate) will start on day -2 and will end on day +30 after stem cell transplant, making the total number of days of drug administration 33 days. Maraviroc will be administered 300mg twice daily orally.
  Interventions: Drug: Maraviroc; Drug: Cyclosporine (in HLA-Unrelated Donor Transplantation); Drug: Tacrolimus (in HLA-Mismatched Related Donor Transplantation); Drug: Methotrexate

INTERVENTIONS:
Drug: Maraviroc — Maraviroc will be administered 300mg twice daily and start on day -2 end on day +30 after stem cell transplant for 33 days.
  Other Names: Selzentry
Drug: Cyclosporine (in HLA-Unrelated Donor Transplantation) — Cyclosporine will be given intravenously at a dose of 2-3 mg/kg starting Day -1. Subsequent dosing will be based on blood levels. Patients were advanced to oral cyclosporine once they could tolerate. The dose should be adjusted accordingly to maintain a suggested target serum level of 150-250 ng/mL. In the absence of aGVHD, the oral cyclosporine dose was reduced by approximately 5% weekly, beginning on or near day 100, and therapy was usually discontinued by Day 180 after transplantation or relapse.
  Other Names: Sandimmune; Gengraf; Neoral
Drug: Tacrolimus (in HLA-Mismatched Related Donor Transplantation) — Tacrolimus will be given orally at a dose of 0.05 mg/kg twince a day or intravenously at a dose of 0.03 mg/kg starting Day -3. Subsequent dosing should be adjusted accordingly to maintain a suggested target serum level of 5-10 ng/mL. Tacrolimus taper can be initiated at a minimum of 100 days post HSCT if there is no evidence of active GVHD. The rate of tapering will be done according institutional practices but patients should be off tacrolimus by Day 180 post HSCT if there is no evidence of active GVHD.
  Other Names: Prograf®; FK506
Drug: Methotrexate — Methotrexate will be administered intravenously at a dose of 15 mg/m^2 on day +1, and 10 mg/m^2 on day +3, +6 and +11 after HSC transplantation.at the doses of 15 mg/m^2 IV bolus on Day +1, and 10 mg/m^2 IV bolus on Days +3, +6 and +11 after hematopoietic stem cell infusion. The Day +11 dose of methotrexate will be not given to those patients who fail to reach white blood cell count (WBC) of more than 1.0×10^9/L.
  Other Names: MTX

SUMMARY:
HLA-mismatched unrelated donor (MMUD) and HLA-haploidentical donor (Haplo Donor) hematopoietic stem cell transplantation (HSCT) is associated with increased graft-versus-host-disease (GVHD) and impaired survival. The chemokine receptor 5 (CCR5) antagonist maraviroc has immunomodulatory properties potentially beneficial for GVHD control as it can blockade lymphocyte chemotaxis without impairing T-cell function. The aim of this study is to evaluate the safety and efficacy of maraviroc combined with standard graft-versus-host-disease prophylaxis in patients with hematologic malignancies after allogeneic stem cell transplantation from HLA-Unrelated or HLA-Mismatched Related donors. Based on the results of our previously small sample study with maraviroc combined with cyclosporine/tacrolimus and methotrexate for prophylaxis of GVHD, the investigators plan to perform the clinical trail.

ELIGIBILITY:
Inclusion Criteria:

1. Age 12-65 years (patient is older than 12.0 and less than 66.0 years old)
2. Patients with acute leukemia, myelodysplastic syndrome or lymphoma who scheduled to undergo allogeneic stem-cell transplantation from HLA-Unrelated or HLA-Mismatched Related donors
3. Renal function: estimated creatinine clearance greater than 40 mL/minute (using the Cockcroft-Gault formula and actual body weight)
4. Hepatic function: Baseline direct bilirubin, alanine aminotransferase (ALT) lower than three times the upper limit of normal
5. Pulmonary disease: forced vital capacity (FVC) or forced expiratory volume at one second (FEV1) > 40% predicted
6. Cardiac ejection fraction > 40%
7. Signed informed consent

Exclusion Criteria:

1. Patients not expected to be available for follow-up in our institution for at least 100 days after the transplant
2. Prior allogeneic transplant
3. Karnofsky Performance Score < 70%
4. Patients who are not undergoing standard GVHD prophylaxis with cyclosporine/tacrolimus and methotrexate
5. Patients with uncontrolled bacterial, viral or fungal infections
6. Patients receiving other investigational drugs for GVHD

Ages: 12 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2014-04; Primary Completion 2016-12 (Estimated); Study Completion 2017-04 (Estimated)

PRIMARY OUTCOMES:
Incidence of Acute GVHD Grades II-IV | 1 Year

SECONDARY OUTCOMES:
Incidence of Acute GVHD Grades III-IV | By day +100 post-HSCT
Incidence of Chronic GVHD | 1 Year
Hematologic Recovery (Neutrophils and Platelets) | Up to day +100 post-HSCT
Disease Relapse or Progression | 1 Year
Incidence of Transplant-Related Mortality | By day +100 post-HSCT
Frequency of Grade 3 or Greater Toxicities | Up to day +100 post-HSCT
Incidence of Grade 2 and 3 Infections | 1 Year
Overall Survival | 1 Year

CONTACTS AND LOCATIONS:
Overall Officials: Hu Chen, M.D., Ph.D., Principal Investigator — Affiliated Hospital to Academy of Military Medical Sciences
Locations (1):
- Department of Hematopoietic Stem Cell Transplantation, Beijing, Beijing Municipality, China